CLINICAL TRIAL: NCT06190886
Title: A First-in-human (FIH), Multicenter, Open-Label, Phase Ia (Dose Escalation)/Phase Ib (Dose Expansion) Study of PTX-912 in Patients with Locally Advanced/Metastatic Solid Tumors
Brief Title: A First-in-human (FIH), Phase I Study of PTX-912 in Patients with Locally Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Proviva Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTX-912-001
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Advanced Cancer; Solid Tumor; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PTX-912 (Experimental): Single or multiple ascending dose of PTX-912
  Interventions: Drug: PTX-912

INTERVENTIONS:
Drug: PTX-912 — Investigation Product Monotherapy

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of escalating doses of PTX-912 in patients with locally advanced or metastatic solid tumors. To evaluate the PK and immunogenicity profile of PTX-912. To evaluate the preliminary anti-tumor activity of PTX-912.

Participants will be treated with PTX-912 via iv infusion, every 2 weeks until progression of disease, unacceptable toxicity, or 12 months of total study therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
2. Male and Female patients age ≥ 18 years on day of signing informed consent.
3. Willing to comply with all protocol-required visits, assessments, and procedures.
4. Patients with locally advanced or metastatic solid tumors who have had disease progression on all available standard of care or for whom no reasonable standard of care exists that would confer clinical benefit.
5. Recovery from all toxicities associated with prior therapy to acceptable baseline status (for laboratory toxicities, see limits for inclusion). NCI CTCAE v5.0 Grade 0 or 1, except for toxicities not considered a safety risk (e.g., alopecia or vitiligo).
6. Measurable disease per RECIST v1.1.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 with no deterioration during Screening.
8. Adequate bone marrow and organ function, defined by the following laboratory results obtained within 14 days before first dose of study drug.
9. Patients with recent major surgery must have adequately recovered with no ongoing complications from the surgery prior to receiving study treatment.
10. Willingness to adhere to the study treatment-specific contraception requirements.
11. Estimated life expectancy of 3 months (12 weeks) or greater as determined by Investigator.

Exclusion Criteria:

1. Has a diagnosis of immunodeficiency.
2. Has an active infection requiring systemic therapy within 4 weeks prior to study treatment.
3. History of or known intolerance, significant hypersensitivity, or anaphylaxis to any components of PTX-912 or any of the excipients.
4. Unresolved toxicities from prior systemic therapy greater than NCI CTCAE grade 1 at time of first dose, except alopecia, vitiligo, and grade 2 neuropathy due to prior chemotherapy.
5. Experienced clinically significant immune-related toxicity from prior immunotherapy that in the opinion of the investigator would preclude protocol therapy or would make the patient inappropriate for the study.
6. Major surgery within 30 days prior to first dose of study drug (with the below exceptions), or anticipation of major surgery during study treatment.
7. Active autoimmune disease requiring systemic treatment within the past 3 months or have a documented history of clinically severe autoimmune disease that requires systemic steroids or immunosuppressive agents.
8. Uncontrolled diabetes mellitus or other uncontrolled immune-related endocrinopathies in the opinion of the investigator.
9. Primary central nervous system (CNS) disease or leptomeningeal disease.
10. Impaired cardiovascular function or clinically significant cardiovascular disease.
11. Abnormal pulmonary function within the previous 6 months, including history of pneumonitis, active pneumonitis, interstitial lung disease requiring the use of steroids, idiopathic pulmonary fibrosis, active pleural effusion, severe dyspnea at rest or requiring supplementary oxygen therapy.
12. History of allogenic, bone marrow, or solid organ transplants.
13. Received a live-virus vaccination ≤14 days prior to first dose of study drug (seasonal flu and other inactivated vaccines that do not contain live virus are permitted).
14. Clinically significant bleeding within 2 weeks prior to first dose of study drug dy.
15. Pregnant or breast-feeding women or expecting to conceive within the projected duration of the trial, starting with the screening visit through 3 months after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
DLTs (dose limiting toxicity) | within 28 days
  Frequency, severity, and duration of treatment-emergent adverse events (TEAEs) and laboratory abnormalities for all dose groups according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0; except for cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) which will be graded according to American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - University of Miami, Miami, Florida
  - Nebraska Cancer Specialists (NCS), Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No